CLINICAL TRIAL: NCT07315295
Title: Maximizing the Benefits of Iron in Ready-to-use Therapeutic Foods for Malnourished Children in Kenya
Acronym: SAMI
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: ETH Zurich (Other)
Responsible Party: Principal Investigator, Nicole Stoffel, Assistantprofessor, ETH Zurich
Allocation: Not Applicable | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: SAMI
Record Dates: First submitted 2025-12-18; First posted 2026-01-02 (Actual); Last update posted 2026-01-02 (Actual); Status verified 2025-12

CONDITIONS: Iron Absorption; Iron Deficiencies; Severly Acutely Malnourished Children; Malnutrition in Children; Anemia
Keywords: Ready to use therapeutic foods (RUFTs); Severe acute malnutrition (SAM); Stable isotopes; Iron bioavailability
MeSH Terms: conditions — Iron Deficiencies; Child Nutrition Disorders; Anemia; Severe Acute Malnutrition | interventions — Therapeutics

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Healthy children (Active Comparator): Healthy children
  Interventions: Other: Iron absorption from RUTF on Day 0
- Children with MAM/SAM (Experimental): children with moderate or severe acute malnutrition
  Interventions: Other: Iron absorption from RUTF on Day 0; Dietary Supplement: Treatment with RUTF for 80 days; Other: Iron absorption from RUTF on Day 20; Other: Iron absorption from RUTF on Day 40; Other: Iron absorption from RUTF on Day 60

INTERVENTIONS:
Other: Iron absorption from RUTF on Day 0 — RUFT with 57Fe
Dietary Supplement: Treatment with RUTF for 80 days — Daily RUTF intake
  Arms: Children with MAM/SAM
Other: Iron absorption from RUTF on Day 20 — RUFT with 57Fe
  Arms: Children with MAM/SAM
Other: Iron absorption from RUTF on Day 40 — RUFT with 57Fe
  Arms: Children with MAM/SAM
Other: Iron absorption from RUTF on Day 60 — RUFT with 57Fe
  Arms: Children with MAM/SAM

SUMMARY:
Reports from the Kenya Red Cross Society (KRCS) in Kwale County, southern Kenya, indicate a limited impact of Ready-to-Use Therapeutic Foods (RUTFs) on malnutrition or anemia. The current RUTF formulation may have an excessively high iron content. In severely acutely malnourished (SAM) children, iron cannot be properly absorbed, leading to life-threatening diarrhea. The overall aim of this project is to develop an improved RUTF treatment that addresses acute malnutrition and anemia in children, ensuring both safety and efficacy. Specifically, to assess the impact of malnutrition on fractional iron absorption (FIA) from RUTFs in children, by comparing healthy children to those with acute malnutrition and by tracking changes in FIA in malnourished children over the course of treatment.

ELIGIBILITY:
Inclusion Criteria:

malnourished children:

* severe acute malnutrition (SAM): WHZ < -3.0
* moderate acute malnutrition (MAM): WHZ < -2.0 a
* treated as outpatients (no acute medical conditions and a positive appetite test)

healthy children:

- healthy: HAZ, WAZ and WHZ = 0

Exclusion Criteria (both groups):

* Hemoglobin ≤7 g/dL
* Presence of acute medical conditions requiring inpatient management

Ages: 12 Months to 54 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 68 (Estimated)
Dates: Start 2025-12-23 (Estimated); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Fractional Iron Absorption | Day 0
Fractional Iron Absorption | Day 20
Fractional Iron Absorption | Day 40
Fractional Iron Absorption | Day 60

SECONDARY OUTCOMES:
Hemoglobin | Day 0
  Iron status parameter
Hemoglobin | Day 20
  Iron status parameter
Hemoglobin | Day 40
  Iron status parameter
Hemoglobin | Day 60
  Iron status parameter
Hemoglobin | Day 80
  Iron status parameter
Serum ferritin | Day 0
  Iron status parameter
Serum Ferritin | Day 20
  Iron status parameter
Serum Ferritin | Day 40
  Iron status parameter
Serum Ferritin | Day 60
  Iron status parameter
soluble transferrin receptor | Day 0
  Iron status parameter
soluble transferrin receptor | Day 20
  Iron status parameter
soluble transferrin receptor | Day 40
  Iron status parameter
soluble transferrin receptor | Day 60
  Iron status parameter
C-reactive protein | Day 0
  inflammation status parameter
C-reactive protein | Day 20
  inflammation status parameter
C-reactive protein | Day 40
  inflammation status parameter
C-reactive protein | Day 60
  inflammation status parameter
α₁-acid glycoprotein | Day 0
  inflammation status parameter
α₁-acid glycoprotein | Day 20
  inflammation status parameter
α₁-acid glycoprotein | Day 40
  inflammation status parameter
α₁-acid glycoprotein | Day 60
  inflammation status parameter
body weight | Day 0
body weight | Day 20
body weight | Day 40
body weight | Day 60
body height | Day 0
body height | Day 20
body height | Day 40
body height | Day 60

CONTACTS AND LOCATIONS:
Locations (2):
- ETH/Oxford/JKUAT research facility, Msambweni, Kwale County, Kenya
- ETH Zurich, Laboratory of Clinical Biopharmacy, Zurich, 8092, Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: No